CLINICAL TRIAL: NCT00152360
Title: The Effect of Xenical on Weight, Risk Factors and Burden of Medication
Brief Title: The Effect of Xenical on Weight and Risk Factors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P03-0151
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2013-04-01 (Estimated); Status verified 2013-03

CONDITIONS: Obesity; Heart Diseases
Keywords: Obesity; weight loss; cardiovascular risk factors; Obesity and obesity related pathology
MeSH Terms: conditions — Obesity; Heart Diseases; Weight Loss | interventions — Orlistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Xenical (Orlistat) (Experimental): Investigating the effectiveness of Xenical on cardiovascular risk factors in the patients of St. Paul's Hospital Lipid Clinic
  Interventions: Drug: Orlistat

INTERVENTIONS:
Drug: Orlistat — See Detailed Description.

SUMMARY:
The purpose of this study is to determine the effect of using the weight loss medication Xenical (generic name - orlistat) on weight loss and change in heart disease risk factors in patients of the Healthy Heart Program Lipid Clinic at St. Paul's Hospital over a three month period. Xenical works by blocking the body's absorption of dietary fat in the gut, allowing it to pass through to be excreted, therefore reducing the intake of fat and calories. This is a pilot study supported by Hoffmann-La Roche Limited which produces Xenical. The aim is to investigate whether weight loss will also result in reductions in heart disease risk factors that may allow for less of a need for medications controlling lipid levels, hypertension and plasma glucose.

DETAILED DESCRIPTION:
Obesity is associated with numerous chronic diseases and increased cardiovascular mortality. It is also an independent risk factor for cardiovascular disease (CVD) in addition to being associated with diabetes and CVD risk factors. Weight loss interventions that target body fat reductions are associated with reductions in cholesterol levels, blood pressure and fasting glucose. Xenical (orlistat) is a gastrointestinal lipase inhibitor which results in a reduction in the absorption of exogenous fat. Studies of up to two years duration have demonstrated that those taking Xenical plus diet lost significantly more weight than those taking placebo plus diet. Coincident with this were decreases in cholesterol levels. The use of Xenical in Type 2 diabetic patients being treated with sulfonylurea resulted in greater discontinuation of the sulfonylurea plus a greater reduction in sulfonylurea dosage compared to placebo. The use of Xenical in the clinical environment has the potential to improve CVD risk factors and potentially reduce the burden of other medications.This is a pilot study to investigate the effectiveness of Xenical on cardiovascular risk factors in the patients of St. Paul's Hospital Lipid Clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index ≥ 27 with one risk factor for cardiovascular disease OR overweight/obese individuals with type 2 diabetes on standard hypoglycemic agents
2. Recently prescribed Xenical at the St. Paul's Hospital Lipid Clinic

Exclusion Criteria:

1. Patients with previous experience using Xenical
2. Patients currently using other weight loss medications.
3. Unable to provide informed consent.
4. Less than 19 years of age

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Weight loss | three months

SECONDARY OUTCOMES:
Lipid profile and insulin, CRP | three months

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Frohlich, MD, Principal Investigator — University of British Columbia
Locations (1):
- Healthy Heart Program/Lipid Clinic, St. Paul's Hospital, Vancouver, British Columbia, Canada